CLINICAL TRIAL: NCT02308020
Title: A Phase 2 Study of Abemaciclib in Patients With Brain Metastases Secondary to Hormone Receptor Positive Breast Cancer, Non-small Cell Lung Cancer, or Melanoma
Brief Title: A Study of Abemaciclib (LY2835219) in Participants With Breast Cancer, Non-small Cell Lung Cancer, or Melanoma That Has Spread to the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15450; I3Y-MC-JPBO (Other: Eli Lilly and Company); 2014-004010-28 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Non-small Cell Lung Cancer; Melanoma; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Brain Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A Abemaciclib: HR+, HER2+ Breast Cancer (Experimental): Abemaciclib 200 milligram (mg) was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or in combination with endocrine therapy (ET). Participants with hormone receptor positive (HR+), HER2+ breast cancer receiving concurrent trastuzumab, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Part B Abemaciclib: HR+, HER2- Breast Cancer (Experimental): Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or for participants in combination with endocrine therapy (ET).
  Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Part C Abemaciclib: Surgical Resection (Experimental): Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or for participants with breast cancer in combination with endocrine therapy (ET). Participants with HR+, HER2+ breast cancer, NSCLC, or melanoma with intracranial lesions for which surgical resection is clinically indicated receiving concurrent trastuzumab, gemcitabine, or pemetrexed, 150 mg abemaciclib was given orally once every 12 hours for 5-14 days prior to surgical resection. Dosing may resume following wound healing on a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Part D Abemaciclib: Non-Small Cell Lung Cancer (NSCLC) (Experimental): Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle. Participants with NSCLC receiving concurrent gemcitabine or pemetrexed, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Part E Abemaciclib: Melanoma (Experimental): Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Part F Abemaciclib: HR+ Breast Cancer, NSCLC, or Melanoma (Experimental): Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or for participants with breast cancer in combination with endocrine therapy (ET). Participants with HR+ (either HER2+ or HER2-) breast cancer, NSCLC, or melanoma and leptomeningeal metastases received concurrent trastuzumab, gemcitabine, or pemetrexed, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of the study drug known as abemaciclib in participants with hormone receptor positive breast cancer, non-small cell lung cancer (NSCLC), or melanoma that has spread to the brain.

ELIGIBILITY:
Inclusion Criteria:

* Have brain metastases secondary to hormone receptor positive breast cancer, NSCLC, or melanoma.
* Have either human epidermal growth factor receptor 2 positive (HER2+) (Study Part A) or negative HER2- (Study Part B) breast cancer.
* Participants in Study Part C must have HR+ breast cancer, NSCLC, or melanoma with brain lesions clinically indicated for surgical resection as well as consent to provide tissue for drug concentration determination after 5 to 14 days of study drug dosing.
* Participants in Part D must have NSCLC of any subtype.
* Participants in Part E must have melanoma of any subtype.
* Participants in Part F must have HR+ breast cancer, NSCLC, or melanoma with leptomeningeal metastases.
* For Parts A, B, D, and E: Must have at least 1 measurable brain lesion ≥10 millimeters (mm) in the longest diameter (LD).
* For Part C (surgical): Have metastatic brain lesion(s) for which surgical resection is clinically indicated.
* Have completed local therapy (surgical resection, whole-breast radiotherapy (WBRT), or SRS) ≥14 days prior to initiating abemaciclib and recovered from all acute effects.
* If receiving concomitant corticosteroids, must be on a stable or decreasing dose for at least 7 days prior to the baseline Gd-MRI.
* Have a Karnofsky performance status of ≥70.
* Have a life expectancy ≥12 weeks.
* For HR+ breast cancer participants in part A, B, C, and F: If currently receiving endocrine therapy, a participant may continue to receive the same endocrine therapy provided that extracranial disease is stable for at least 3 months and central nervous system (CNS) disease progression has occurred while on this endocrine therapy. If these conditions are not met, participants must discontinue endocrine therapy prior to initiation of abemaciclib.
* For HER2+ breast cancer participants in parts A, C, and F: participants may receive concurrent treatment (ongoing or initiated simultaneously with abemaciclib) with IV trastuzumab.
* For NSCLC participants in parts C, D, and F: if currently receiving gemcitabine or pemetrexed (single-agent or in combination with another therapy), a participant may continue to receive 1 of these 2 therapies provided that extracranial disease is stable for at least 6 weeks and CNS disease progression has occurred while on this therapy.
* Have adequate organ function.

Exclusion Criteria:

* Require immediate local therapy, including but not limited to WBRT, SRS, or surgical resection, for treatment of brain metastases.
* Are taking concurrent enzyme-inducing antiepileptic drugs (EIAED).
* Have evidence of significant (ie, symptomatic) intracranial hemorrhage.
* For Parts A, B, C, D, E: Have evidence of leptomeningeal metastases. Note: discrete dural metastases are permitted.
* Have experienced >2 seizures within 4 weeks prior to study entry.
* For Parts A, B, D, E, and F: Have previously received treatment with any cyclin dependent kinase 6 (CDK6) inhibitor. For Part C participants may have received prior palbociclib or ribociclib, but not abemaciclib treatment.
* Have known contraindication to Gd-MRI.
* Have a preexisting chronic condition resulting in persistent diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-459) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (43):
- United States (19):
  - City of Hope National Medical Center, Duarte, California
  - University of California - San Diego, La Jolla, California
  - Univ of California San Francisco, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Kaiser Permanente Center for Health Research, Honolulu, Hawaii
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Providence Health and Services, Portland, Oregon
  - SMO Sarah Cannon Research Inst., Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newcastle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southport
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Belgium (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa, Canada
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Brieuc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Israel (2):
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Tolaney SM, Sahebjam S, Le Rhun E, Bachelot T, Kabos P, Awada A, Yardley D, Chan A, Conte P, Dieras V, Lin NU, Bear M, Chapman SC, Yang Z, Chen Y, Anders CK. A Phase II Study of Abemaciclib in Patients with Brain Metastases Secondary to Hormone Receptor-Positive Breast Cancer. Clin Cancer Res. 2020 Oct 15;26(20):5310-5319. doi: 10.1158/1078-0432.CCR-20-1764. Epub 2020 Jul 21. PMID 32694159
- See also: Click here for more information about this study: A Study of Abemaciclib (LY2835219) in Participants With Breast Cancer, Non-small Cell Lung Cancer, or Melanoma that has Spread to the Brain — https://lillytrialguide.com/en-US/studies/advanced-cancer/JPBO#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who died or discontinued study treatment due to progressive disease and is in follow up.
Groups:
- Part A Abemaciclib: Hormone Receptor (HR+) HER2+ Breast Cancer: Abemaciclib 200 milligram (mg) was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or in combination with endocrine therapy (ET). Participants with hormone receptor positive (HR+), hormone epidermal growth factor receptor 2 positive (HER2+) breast cancer receiving concurrent trastuzumab, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part B Abemaciclib: HR+, HER2- Breast Cancer: Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or in combination with endocrine therapy (ET).
  Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Part A Abemaciclib: Hormone Receptor (HR+) HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part C Abemaciclib: Surgical Resection | Part D Abemaciclib: Non-Small Cell Lung Cancer (NSCLC) | Part E Abemaciclib: Melanoma | Part F Abemaciclib: HR+ Breast Cancer, NSCLC, or Melanoma
Started | 27 | 58 | 9 | 28 | 23 | 17
Received at Least One Dose of Study Drug | 27 | 58 | 9 | 28 | 23 | 17
Completed | 23 | 38 | 6 | 24 | 19 | 12
Not Completed | 4 | 20 | 3 | 4 | 4 | 5
Not completed — Lost to Follow-up | 1 | 7 | 0 | 0 | 1 | 2
Not completed — Sponsor Decision | 0 | 8 | 0 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 3 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A Abemaciclib: HR+, HER2+ Breast Cancer: Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or in combination with endocrine therapy (ET). Participants with hormone receptor positive HR+, HER2+ breast cancer receiving concurrent trastuzumab, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D Abemaciclib: NSCLC: Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle. Participants with NSCLC receiving concurrent gemcitabine or pemetrexed, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Total: Total of all reporting groups
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part C Abemaciclib: Surgical Resection | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma | Part F Abemaciclib: HR+ Breast Cancer, NSCLC, or Melanoma | Total
Number analyzed (Participants) | 27 | 58 | 9 | 28 | 23 | 17 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (10.9) | 54.1 (10.5) | 57.0 (17.9) | 58.4 (10.9) | 55.1 (14.4) | 50.1 (12.3) | 54.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 57 | 8 | 14 | 11 | 14 | 131
  Male | 0 | 1 | 1 | 14 | 12 | 3 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 21 | 42 | 8 | 20 | 20 | 14 | 125
  Unknown or Not Reported | 6 | 13 | 1 | 8 | 2 | 2 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 1 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 0 | 1 | 0 | 1 | 7
  White | 17 | 35 | 7 | 20 | 22 | 14 | 115
  More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 7 | 15 | 1 | 7 | 1 | 2 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Austria | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Belgium | 4 | 8 | 0 | 3 | 3 | 0 | 18
  United States | 11 | 24 | 7 | 12 | 7 | 10 | 71
  Italy | 0 | 4 | 0 | 2 | 9 | 0 | 15
  Israel | 1 | 2 | 0 | 1 | 1 | 1 | 6
  Australia | 2 | 2 | 1 | 2 | 1 | 1 | 9
  France | 7 | 14 | 1 | 7 | 1 | 2 | 32
  Spain | 2 | 2 | 0 | 1 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR): Objective Intracranial Response Rate (OIRR)
Description: OIRR is the percentage of participants with a (CR) or (PR) based on the Response Assessment in Neuro-Oncology Brain Metastasis (RANO-BM) response criteria. CR is measurable target lesions, the disappearance of all central nervous system (CNS) target lesions for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically. PR is at least a 30% decrease in the sum longest duration (LD) of CNS target lesions, taking as reference the baseline sum LD for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. Nontarget lesions requires disappearance CNS non-target lesions and no new CNS lesions. Stable disease (SD) is less than (<)30% decrease relative to baseline but <20% increase in sum LD relative to nadir. Progressive disease (PD) is greater than or equal to (≥) 20% increase in sum LD relative to nadir and a relative increase of 20%, ≥1 lesion must increase by absolute value of ≥5 millimeter (mm).
Time Frame: Baseline to Objective Disease Progression (Up to 36 Months)
Population: All participants who had evaluable OIRR data with at least one measurable brain lesion at baseline (per RANO-BM) and for whom at least one post-baseline overall response assessment for intracranial disease is available. Parts C and F were exploratory per protocol.
Measure: Number; unit: percentage of participants
Groups:
- Part B Abemaciclib: HR+, HER2- Breast Cancer: Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or for in combination with endocrine therapy (ET).
  Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 23 | 52 | 23 | 22
percentage of participants | 0 | 5.8 | 0 | 0

2. Secondary Outcome: Percentage of Participants With CR, PR, Stable Disease (SD), Progressive Disease (PD), or Not Evaluable (NE): Best Overall Intracranial Response (BOIR)
Description: Percentage of Participants with BOIR was categorized as CR, PR, SD, PD or NE, as defined by RANO-BM, from baseline until the earliest of objective progression according to brain metastases response criteria or start of new anticancer therapy. CR is measurable target lesions, the disappearance of all CNS target lesions for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically. PR is at least a 30% decrease in the sum LD of CNS target lesions, taking as reference the baseline sum LD for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. SD is <30% decrease relative to baseline but <20% increase in sum LD relative to nadir. PD is greater than or equal to (≥) 20% increase in sum LD relative to nadir and a relative increase of 20%, ≥1 lesion must increase by absolute value of ≥5 mm. NE is absent (no abnormality; normal), or non-evaluable (NE).
Time Frame: Baseline to Earliest Objective Progression or Start of New Anticancer Therapy (Up to 36 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 23 | 52 | 23 | 22
percentage of participants
  Partial Response | 0 | 5.8 | 0 | 0
  Stable Disease | 52.2 | 65.4 | 43.5 | 31.8
  Progressive Disease | 47.8 | 28.8 | 56.5 | 68.2
  Not Evaluable | 0 | 0 | 0 | 0

3. Secondary Outcome: Duration of CR or PR: Duration of Intracranial Response (DOIR)
Description: DOIR is measured from the date of first evidence of a confirmed response (CR or PR), as defined by RANO-BM, to the date objective progression or death from any cause. CR is measurable target lesions, the disappearance of all CNS target lesions for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically. PR is at least a 30% decrease in the sum LD of CNS target lesions, taking as reference the baseline sum LD for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. Participants who have neither progressed nor died were censored on the day of their last radiographic tumor assessment or on the date of response. PD is greater than or equal to (≥) 20% increase in sum LD relative to nadir and a relative increase of 20%, ≥1 lesion must increase by absolute value of ≥5 mm. DOIR was summarized using Kaplan-Meier estimates.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death from Any Cause (Up to 36 Months)
Population: All participants who had a confirmed intracranial response of CR or PR (per RANO-BM) and for whom at least one post-baseline overall intracranial response with a measurable duration is available. Parts C and F were exploratory per protocol.
Measure: Median (Full Range); unit: Months
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 0 | 3 | 0 | 0
Months |  | 8.8 [3.0 to 14.3] |  |

4. Secondary Outcome: Percentage of Participants With Best Overall Intracranial Response (BOIR) of CR, PR, or SD: Intracranial Disease Control Rate (IDCR)
Description: Percentage of participants with BOIR of CR, PR, or SD: IDCR, as defined by RANO-BM is reported. CR is measurable target lesions, the disappearance of all central nervous system CNS target lesions for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically. PR is at least a 30% decrease in the sum LD of CNS target lesions, taking as reference the baseline sum LD for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. Nontarget lesions requires disappearance CNS non-target lesions and no new CNS lesions. SD is less than (<)30% decrease relative to baseline but <20% increase in sum LD relative to nadir. PD is greater than or equal to (≥) 20% increase in sum LD relative to nadir and a relative increase of 20%, ≥1 lesion must increase by absolute value of ≥5 mm.
Time Frame: Baseline to Disease Progression or Start of New Anticancer Therapy (Up to 36 Months)
Population: All participants who had evaluable OIRR data with at least one measurable brain lesion at baseline (per RANO-BM) and for whom at least one post-baseline overall response assessment. Parts C and F were exploratory per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 23 | 52 | 23 | 22
percentage of participants | 52.2 | 71.2 | 43.5 | 31.8

5. Secondary Outcome: Percentage of Participants With BOIR of CR, PR, or SD With Duration of SD for at Least 6 Months: Intracranial Clinical Benefit Rate (ICBR)
Description: ICBR is the percentage of participants with BOIR of CR, PR, or SD with duration of SD for at least 6 months, as defined by RANO-BM. CR is measurable target lesions, the disappearance of all CNS target lesions for at least 4 weeks; no new lesions; no corticosteroids; stable or improved clinically. PR is at least a 30% decrease in the sum LD of CNS target lesions, taking as reference the baseline sum LD for at least 4 weeks; no new lesions; stable to decreased corticosteroid dose; stable or improved clinically. SD is <30% decrease relative to baseline but <20% increase in sum LD relative to nadir. PD is greater than or equal to (≥) 20% increase in sum LD relative to nadir and a relative increase of 20%, ≥1 lesion must increase by absolute value of ≥5 mm.
Time Frame: Baseline to Disease Progression or Start of New Anticancer Therapy (Up to 36 Months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 23 | 52 | 23 | 22
percentage of participants | 13.0 | 26.9 | 26.1 | 9.1

6. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from baseline to the date of death from any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for a particular analysis, OS was censored for that analysis at the date of last contact prior to the data inclusion cutoff date (contacts considered in the determination of last contact date include adverse event (AE) date, tumor assessment date, visit date, and last known alive date). OS was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to the Date of Death from Any Cause (Up to 5 Years)
Population: All participants who received at least one dose of study drug. Parts C and F were exploratory per protocol. Censored participants in Part A = 4, Part B = 20, Part D = 4, Part E = 4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 27 | 58 | 28 | 23
months | 10.06 [4.21 to 14.30] | 13.38 [9.60 to 20.84] | 7.13 [3.65 to 9.37] | 2.93 [1.22 to 4.31]

7. Secondary Outcome: Percentage of Participants With a Best Response of CR or PR: Extracranial Objective Response Rate (EORR)
Description: The percentage of participants with a best response of CR or PR objective response rate is complete response (CR) + partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. PD is defined as at least a 20% increase in the sum LD of CNS target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) and the 20% increase must be at least one lesion must increase by an absolute value of ≥5 mm to be considered progression.
Time Frame: Baseline to Disease Progression (Up to 36 Months)
Population: All participants who received at least one dose of study drug. Parts C and F were exploratory per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 27 | 58 | 28 | 23
percentage of participants | 0 | 1.7 | 3.6 | 0

8. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR, PR, or SD: Extracranial Disease Control Rate (EDCR)
Description: Disease control rate (DCR) (CR+ PR+ SD) per RECIST v1.1. is defined as the percentage of participants with best overall response of CR, PR, or SD. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions. PD is defined as at least a 20% increase in the sum LD of CNS target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) and the 20% increase must be at least one lesion must increase by an absolute value of ≥5 mm to be considered progression.
Time Frame: Baseline to Disease Progression or Start of New Anticancer Therapy (Up to 36 Months)
Population: All participants who received at least one dose of study drug. Parts C and F were exploratory per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 27 | 58 | 28 | 23
percentage of participants | 40.7 | 51.7 | 39.3 | 26.1

9. Secondary Outcome: Progression Free Survival (PFS) Bi-compartmental
Description: PFS was measured from baseline to objective progression (intracranial or extracranial) as defined by (RANO-BM.) or death from any cause. Participants who have neither progressed nor died were censored at the day of their last radiographic tumor assessment. PD is greater than or equal to (≥) 20% increase in sum LD relative to nadir and a relative increase of 20%, ≥1 lesion must increase by absolute value of ≥5 mm. PFS was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Objective Disease Progression or Death from Any Cause (Up to 36 Months)
Population: All participants who received at least one dose of study drug. Censored participants Part A = 1, Part B =2, Part D = 1 and Part E = 1. Parts C and F were exploratory per protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 27 | 58 | 28 | 23
Months | 2.07 [1.35 to 3.32] | 4.41 [2.60 to 5.46] | 1.45 [1.35 to 2.76] | 1.22 [1.02 to 1.55]

10. Secondary Outcome: Change From Baseline in Neurologic Symptoms on the MD Anderson Inventory-Brain Tumor (MDASI-BT) Subscale
Description: The MDASI-BT is an instrument to assess multi-symptoms in participants with brain tumor metastases (including those with brain metastases secondary to breast cancer). The MDASI-BT of participants with a change from baseline is reported as mean core symptoms, mean brain tumor symptoms, and symptom groupings (mean focal neurologic deficit, mean generalized/disease status symptoms, and mean gastrointestinal symptoms). The mean of all symptom subscale items was calculated where 0 equals "not present" and 10 equals "as bad as you can imagine." A change from baseline with negative values indicate improvement, positive values indicate worsening.
Time Frame: Baseline, Cycle 3 (Up to 63 Days)
Population: All participants who received at least one dose of study drug and had at least 1 baseline and an evaluable post baseline assessment. Parts C and F were exploratory per protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Part A Abemaciclib: HR+, HER2+ Breast Cancer: Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or for in combination with endocrine therapy (ET). Participants with hormone receptor positive HR+, HER2+ breast cancer receiving concurrent trastuzumab, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma
Number analyzed (Participants) | 11 | 35 | 10 | 7
units on a scale
  mean core symptom severity | -0.98 (0.86) | -0.17 (0.99) | -0.38 (1.19) | -0.53 (0.62)
  mean brain tumor symptom severity: number analyzed (Participants) | 11 | 35 | 9 | 7
  mean brain tumor symptom severity | -0.47 (0.57) | -0.29 (1.05) | -0.10 (1.22) | 0.31 (1.11)
  mean focal neurologic deficit symptom severity: number analyzed (Participants) | 11 | 35 | 9 | 7
  mean focal neurologic deficit symptom severity | -0.84 (0.92) | -0.36 (1.23) | -0.44 (0.58) | 0.54 (1.16)
  mean generalized disease status: number analyzed (Participants) | 11 | 35 | 9 | 7
  mean generalized disease status | -0.47 (1.03) | 0 (1.39) | 0.28 (1.51) | 0.01 (0.89)
  mean gastrointestinal symptom: number analyzed (Participants) | 10 | 34 | 8 | 7
  mean gastrointestinal symptom | -1.35 (2.11) | 0.40 (1.91) | 1.00 (1.46) | 0 (0.29)

11. Secondary Outcome: Pharmacokinetics (PK): Steady State Minimum Concentration (Cmin) of Abemaciclib and Its Metabolites LSN2839567 (M2), LSN3106726 (M20), and LSN3106729 (M18)
Description: A PK plasma sample was taken prior to abemaciclib dose to analyze the minimum concentrations of abemaciclib and its metabolites (Cmin) - Individual Cmin values were averaged if there were 3 or more available data points, otherwise individual data are reported.
Time Frame: Parts A, B, D, E, F, Cycle 3, Day 1: Predose; Part C, Cycle 4, Day 1: Predose
Population: All participants who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Part A 150 mg Abemaciclib: HR+, HER2+ Breast Cancer: Participants with HR+, HER2+ breast cancer received 150 mg abemaciclib orally once every 12 hours on days 1-21 of a 21-day cycle.
- Part B 200 mg Abemaciclib: HR+, HER2- Breast Cancer: Participants with HR+, HER2- breast cancer received 200 mg abemaciclib given orally once every 12 hours on days 1-21 of a 21-day cycle.
- Part C 200 mg Abemaciclib: Surgical Resection: Participants with HR+ breast cancer, NSCLC, or melanoma with intracranial lesions for which surgical resection is clinically indicated received 200 mg abemaciclib given orally once every 12 hours for 5-14 days prior to surgical resection.
- Part D 200 mg Abemaciclib: NSCLC: Participants with NSCLC received 200 mg abemaciclib given orally once every 12 hours on days 1-21 of a 21-day cycle.
- Part E 200 mg Abemaciclib: Melanoma: Participants with melanoma received 200 mg abemaciclib given orally once every 12 hours on days 1-21 of a 21-day cycle.
- Part F 200 mg Abemaciclib: HR+ Breast Cancer, NSCLC, Melanoma: Participants with HR+ (either HER2+ or HER2-) breast cancer, NSCLC, or melanoma and leptomeningeal metastases received 200 mg abemaciclib given orally once every 12 hours on days 1-21 of a 21-day cycle.
Arm/Group | Part A 150 mg Abemaciclib: HR+, HER2+ Breast Cancer | Part B 200 mg Abemaciclib: HR+, HER2- Breast Cancer | Part C 200 mg Abemaciclib: Surgical Resection | Part D 200 mg Abemaciclib: NSCLC | Part E 200 mg Abemaciclib: Melanoma | Part F 200 mg Abemaciclib: HR+ Breast Cancer, NSCLC, Melanoma
Number analyzed (Participants) | 3 | 12 | 1 | 5 | 2 | 4
nanogram/milliliter (ng/mL)
  Abemaciclib | 133 (13.4) | 120 (186) | NA (NA) — N=1, Geometric mean and coefficient of variation (CV) were not calculated. Individual value reported: 256 ng/mL | 306 (33.5) | NA (NA) — N=2, Geometric mean and CV were not calculated. Individual values reported: 99.7 ng/mL and 222 ng/mL | 142 (80.0)
  LSN2839567 (M2) | 72.6 (8.23) | 77.3 (121) | NA (NA) — N=1, Geometric mean and CV were not calculated. Individual value reported: 98.8 ng/mL | 100 (77.5) | NA (NA) — N=2, Geometric mean and CV were not calculated. Individual values reported: 61.6 ng/mL and 90.7 ng/mL | 68.5 (150)
  LSN3106726 (M20) | 158 (25.0) | 133 (160) | NA (NA) — N=1, Geometric mean and CV were not calculated. Individual value reported: 181 ng/mL | 203 (43.3) | NA (NA) — N=2, Geometric mean and CV were not calculated. Individual values reported: 109 ng/mL and 172 ng/mL | 122 (137)
  LSN3106729 (M18): number analyzed (Participants) | 3 | 11 | 1 | 5 | 2 | 4
  LSN3106729 (M18) | 36.8 (39.3) | 42.4 (85.6) | NA (NA) — N=1, Geometric mean and CV were not calculated. Individual value reported: 28.2 ng/mL | 28.9 (108) | NA (NA) — N=2, Geometric mean and CV were not calculated. Individual values reported: 22.2 ng/mL and 44.2 ng/mL | 27.0 (242)

ADVERSE EVENTS:
Time Frame: Up to 36 Months
Description: All participants who received at least one dose of study drug.
Groups:
- Part F: Abemaciclib HR+ Breast Cancer, NSCLC, or Melanoma: Abemaciclib 200 mg was administered orally once every 12 hours on days 1-21 of a 21-day cycle when administered as a single agent or for participants with breast cancer in combination with Endocrine Therapy (ET). Participants with HR+ (either HER2+ or HER2-) breast cancer, NSCLC, or melanoma and leptomeningeal metastases received concurrent trastuzumab, gemcitabine, or pemetrexed, 150 mg abemaciclib was given orally once every 12 hours on days 1-21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A Abemaciclib: HR+, HER2+ Breast Cancer | Part B Abemaciclib: HR+, HER2- Breast Cancer | Part C Abemaciclib: Surgical Resection | Part D Abemaciclib: NSCLC | Part E Abemaciclib: Melanoma | Part F: Abemaciclib HR+ Breast Cancer, NSCLC, or Melanoma
All-Cause Mortality (participants affected / at risk) | 23/27 | 38/58 | 6/9 | 24/28 | 19/23 | 12/17
Serious Adverse Events (participants affected / at risk) | 6/27 | 16/58 | 3/9 | 8/28 | 4/23 | 7/17
Other Adverse Events (participants affected / at risk) | 23/27 | 55/58 | 8/9 | 27/28 | 16/23 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Abemaciclib: HR+, HER2+ Breast Cancer (N=27) | Part B Abemaciclib: HR+, HER2- Breast Cancer (N=58) | Part C Abemaciclib: Surgical Resection (N=9) | Part D Abemaciclib: NSCLC (N=28) | Part E Abemaciclib: Melanoma (N=23) | Part F: Abemaciclib HR+ Breast Cancer, NSCLC, or Melanoma (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shunt infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Abemaciclib: HR+, HER2+ Breast Cancer (N=27) | Part B Abemaciclib: HR+, HER2- Breast Cancer (N=58) | Part C Abemaciclib: Surgical Resection (N=9) | Part D Abemaciclib: NSCLC (N=28) | Part E Abemaciclib: Melanoma (N=23) | Part F: Abemaciclib HR+ Breast Cancer, NSCLC, or Melanoma (N=17)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 12 (14) | 4 (7) | 5 (6) | 2 (5) | 5 (5)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 7 (10) | 4 (6) | 4 (6) | 3 (5) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (9) | 3 (8) | 4 (7) | 1 (2) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 6 (8) | 17 (32) | 4 (6) | 7 (9) | 5 (8) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 11 (12) | 4 (5) | 8 (11) | 3 (4) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 9 (14) | 2 (4) | 2 (2) | 5 (5) | 4 (4)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 9 (11) | 0 (0) | 7 (7) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 15 (26) | 45 (100) | 4 (6) | 15 (21) | 5 (6) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (11) | 26 (32) | 2 (2) | 8 (10) | 1 (1) | 7 (10)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8) | 20 (31) | 2 (2) | 4 (4) | 1 (1) | 5 (6)
Chills (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (9) | 28 (31) | 2 (2) | 11 (16) | 4 (4) | 9 (9)
Gait disturbance (General disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (6) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (4) | 6 (7) | 2 (4) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 3 (4) | 2 (5) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 5 (6) | 1 (1) | 2 (4) | 2 (3) | 1 (2)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 6 (6) | 2 (2) | 4 (5) | 1 (2) | 2 (2)
Weight increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 19 (19) | 2 (2) | 7 (10) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 6 (6) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (9) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7) | 11 (17) | 2 (5) | 2 (2) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 1 (2) | 2 (9) | 1 (1) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 3 (3) | 1 (1) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (5) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 14 (23) | 2 (3) | 4 (4) | 2 (3) | 3 (3)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 3 (3) | 12 (19) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 4 (5) | 3 (3) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (2) | 2 (2) | 5 (8) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (9) | 1 (2) | 5 (5) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: Protocol (2014-11-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02308020/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT02308020/SAP_001.pdf
  • Study Protocol: Protocol Amendment (d) (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT02308020/Prot_002.pdf